CLINICAL TRIAL: NCT01313390
Title: DORA: A Phase I and Randomized Phase II Study of Docetaxel and RAD001 (Everolimus) in Advanced/Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Everolimus and Docetaxel in Treating Patients With Recurrent, Locally Advanced, or Metastatic Head and Neck Cancer
Acronym: DORA
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000696702; CRUK-UCL-06/053; EU-20959; ISRCTN-73814534; EUDRACT-2007-001951-20; CRUK-UCL-CTA-20363/0229/011-00; NOVARTIS-CRUK-UCL-06/053; AVENTIS-CRUK-UCL-06/053
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent verrucous carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; recurrent squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; salivary gland squamous cell carcinoma; stage III salivary gland cancer; stage IV salivary gland cancer; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms; Tongue Neoplasms | interventions — Docetaxel; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: docetaxel
Drug: everolimus
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving everolimus together with docetaxel is more effective than giving docetaxel alone in treating patients with head and neck cancer.

PURPOSE: This phase I/II trial is studying the side effects and best dose of everolimus given together with docetaxel in treating patients with recurrent, locally advanced, or metastatic head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the safety and tolerability of the combination of everolimus and docetaxel in treating patients with recurrent, locally advanced or metastatic squamous cell carcinoma of the head and neck. (Phase I)
* To determine the maximum-tolerated dose and recommended phase II dose of everolimus when combined with docetaxel in these patients. (Phase I)
* To examine the response rates in patients receiving the combination of docetaxel and everolimus and those receiving docetaxel alone. (Phase II)

Secondary

* To investigate possible pharmacokinetic interactions between docetaxel and everolimus in these patients. (Phase I)
* To investigate the effect of everolimus on downstream targets of mTOR in tumor in these patients. (Phase I)
* To examine the time to progression after docetaxel and everolimus in these patients. (Phase II)
* To perform a pilot study to attempt to identify predictors of response, including evaluation of EGFR family member expression, mutations, or amplifications. (Phase II)
* To attempt to identify downstream targets of the EGFR pathway including phosphorylation of S6 and phosphorylation of AKT. (Phase II)

OUTLINE: This is a multicenter, phase I, dose-escalation study of everolimus with docetaxel followed by a randomized phase II study.

* Phase I: Patients receive docetaxel IV over 1 hour on day 1 and escalating doses of oral everolimus on days 1, 8, and 15. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 courses of therapy, patients may continue to receive everolimus weekly as a single agent until evidence of progressive disease.
* Phase II: Patients are randomized to 1 of 2 treatment arms:

  * Arm A: Patients receive docetaxel IV over 1 hour on day 1.Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients with progressive disease are eligible to cross over into the everolimus arm at the investigator's discretion.
  * Arm B: Patients receive docetaxel as in arm A and oral everolimus (at a dose determined in the phase I portion of the study) on days 1, 8, and 15. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. After the completion of combination therapy, patients may continue to receive maintenance everolimus weekly, at the investigator's discretion.

Blood samples are collected for pharmacokinetic monitoring in the phase I study. Tissue samples are collected at baseline and periodically during the study for biomarker and other laboratory analysis.

After completion of study treatment, patients are followed up every 3 months for at least 1 year.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

PROJECTED ACCRUAL: Approximately 18 patients will be accrued for phase I and a total of 100 patients will be accrued for phase II of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck

  * Locally advanced or metastatic disease

    * No patients with locally advanced disease for whom radiotherapy is indicated
  * Recurrent disease
  * Incurable disease
* Measurable disease by RECIST criteria

  * Recurrent disease within a prior radiation field can be considered to be measurable
* Patients may have received 1 line of prior chemotherapy (but not a taxane) for locally advanced or metastatic disease
* Patients may have received prior radiation therapy for locally advanced or metastatic disease (but must have completed the radiotherapy > 6 months before recruitment)

  * No disease relapsed within 6 months of radiotherapy
* No evidence of central nervous system metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 12 weeks
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* Urea and creatinine normal
* Serum bilirubin normal
* AST or ALT ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase < 2.5 times ULN
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months (female) or 2 months (male) after the last dose of the study treatment
* No uncontrolled infection
* No mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study
* No prior malignancy likely to interfere with the patient's ability to comply with treatment and/or follow up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy for any cancer, except for head and neck cancer
* No prior taxane
* No prior therapy with any erbB inhibitors (except cetuximab given with radiotherapy, as indicated in treatment algorithm)
* More than 6 months since prior radiotherapy for locally advanced or metastatic disease
* At least 4 weeks since prior investigational drug
* No concurrent use of drugs known to inhibit CYP3A4 (except dexamethasone), or block P-glycoprotein, including grapefruit juice
* No other concurrent chemotherapy, immunotherapy, hormonal cancer therapy, radiotherapy, or experimental medications
* No concurrent live vaccines during everolimus therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose and recommended phase II dose of everolimus in combination with docetaxel (phase I)
Safety and tolerability of the combination of everolimus and docetaxel
Response using RECIST criteria (phase II)

SECONDARY OUTCOMES:
Pharmacokinetic profile of docetaxel with and without concurrent everolimus (phase I)
Pharmacokinetic profile of everolimus with and without concurrent docetaxel (phase I)
Time to progression following response (time from treatment start to tumor progression as defined by RECIST criteria) (phase II)
Mutations in EGFR1, AKT, mTOR, ras, or p53 to be tested on paraffin-embedded tissue from the primary or secondary tumor; results to be correlated with outcome (phase II)
Amplifications of EGFR1 and bcl2 expression to be tested by FISH and immunostaining on paraffin-embedded tissue from primary tumor; results to be correlated with outcome (phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Boshoff, Principal Investigator — University College London (UCL) Cancer Institute
Locations (1):
- UCL Cancer Institute, London, England, United Kingdom